CLINICAL TRIAL: NCT03114644
Title: Reading Stories to Premature Babies Reinforces Mother-baby Synchronies?
Acronym: SynchroPrema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2014_843_0010
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Premature Infant; Mother-Baby Synchrony
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Babies born prematurely between 27 and 37 SA (Other)
  Interventions: Other: Physiologically evaluate the impact of reading history on the mother-baby synchronies in a context of premature birth requiring hospitalization in neonatal medicine.

INTERVENTIONS:
Other: Physiologically evaluate the impact of reading history on the mother-baby synchronies in a context of premature birth requiring hospitalization in neonatal medicine. — Physiologically evaluate the impact of reading history on the mother-baby synchronies in a context of premature birth requiring hospitalization in neonatal medicine.

SUMMARY:
Observations of the early interactions between the infant and his parents highlighted the existence of rhythmic and reciprocal communications that serve as a basis for the mother-baby relationship and the emotional and cognitive development of the baby.

DETAILED DESCRIPTION:
Observations of the early interactions between the infant and his parents highlighted the existence of rhythmic and reciprocal communications that serve as a basis for the mother-baby relationship and the emotional and cognitive development of the baby. In this study, the investigator proposes to focus on premature births (before 37 years) because prematurity disrupts the synchronization of these mother-baby communication. For several years, reading of stories and nursery rhymes has been used by the liaison child psychiatry team in the neonatal medicine and pediatric intensive care unit of the University Hospital of Amiens, as a therapeutic mediation tool allowing And support for parent-child interactions. Thus, it is desirable to explore the impact of reading stories and rhymes on mother-baby synchronies. The study is innovative because it simultaneously explores several fields: physiological, neuroendocrine, cognitive and psychic. A pilot study carried out in 2013 showed the feasibility of this exploration in the three protagonists of the interaction: mother, preterm baby and reader.

ELIGIBILITY:
Inclusion Criteria:

* A premature birth between 27 and 37 SA
* At the time of the transfers, the latter must be hospitalized in intensive care and extubated

Exclusion Criteria:

For the baby:

* an unstable medical condition
* Serious somatic complications
* genetic or neurological diseases
* a twin.

For the mother:

* an impossibility to understand and speak the French language
* a mental or cognitive pathology
* an addiction to alcohol or other psychoactive substances
* persons under guardianship or curatorship or deprived of their liberty by a judicial or administrative decision

Ages: 25 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-01-17 (Actual); Primary Completion 2024-01-17 (Estimated); Study Completion 2024-01-17 (Estimated)

PRIMARY OUTCOMES:
Analysis of cardio-respiratory synchronies and vagal tone | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France